CLINICAL TRIAL: NCT02990000
Title: Enhancing Mental Health Care by Scientifically Matching Patients to Providers' Strengths
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); University at Albany (Other); Psychological and Behavioral Consultants (Other); Outcome Referrals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IHS-1503-28573
Record Dates: First submitted 2016-11-29; First posted 2016-12-12 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-05

CONDITIONS: Mental Illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pragmatic Match (No Intervention): Randomly assigned, by a case-assigning administrator, to naturalistic treatment with a pragmatically matched provider (control group)
- Scientific Match (Experimental): Randomly assigned, by a case-assigning administrator, to naturalistic treatment with a scientifically matched provider (experimental group)
  Interventions: Behavioral: Scientific Match

INTERVENTIONS:
Behavioral: Scientific Match — We have developed an innovative, personalized Match System based on provider track records determined with a multidimensional outcomes tool - the Treatment Outcome Package (TOP). Specifically, patients are assigned to therapists with previously established strengths (i.e., being historically effective) in treating their primary problems (e.g., depression, anxiety).
  Other Names: Match System
  Arms: Scientific Match

SUMMARY:
Research has shown that mental health care (MHC) providers differ significantly in their ability to help patients. In addition, providers demonstrate different patterns of effectiveness across symptom and functioning domains. For example, some providers are reliably effective in treating numerous patients and problem domains, others are reliably effective in some domains (e.g., depression, substance abuse) yet appear to struggle in others (e.g., anxiety, social functioning), and some are reliably ineffective, or even harmful, across patients and domains. Knowledge of these provider differences is based largely on patient-reported outcomes collected in routine MHC settings.

Unfortunately, provider performance information is not systematically used to refer or assign a particular patient to a scientifically based best-matched provider. MHC systems continue to rely on random or purely pragmatic case assignment and referral, which significantly "waters down" the odds of a patient being assigned/referred to a high performing provider in the patient's area(s) of need, and increases the risk of being assigned/referred to a provider who may have a track record of ineffectiveness. This research aims to solve the existing non-patient-centered provider-matching problem.

Specifically, the investigators aim to demonstrate the comparative effectiveness of a scientifically-based patient-provider match system compared to status quo pragmatic case assignment. The investigators expect in the scientific match group significantly better treatment outcomes (e.g., symptoms, quality of life) and higher patient satisfaction with treatment. The investigators also expect to demonstrate feasibility of implementing a scientific match process in a community MHC system and broad dissemination of the easily replicated scientific match technology in diverse health care settings. The importance of this work for patients cannot be understated. Far too many patients struggle to find the right provider, which unnecessarily prolongs suffering and promotes health care system inefficiency. A scientific match system based on routine outcome data uses patient-generated information to direct this patient to this provider in this setting. In addition, when based on multidimensional assessment, it allows a wide variety of patient-centered outcomes to be represented (e.g., symptom domains, functioning domains, quality of life).

DETAILED DESCRIPTION:
Background and Significance:

Mental illness is an extraordinary and highly burdensome public health problem. Unfortunately, even for individuals who access mental health care (MHC), the care is too often substandard. Research has consistently demonstrated that approximately 10-15% of patients will deteriorate or experience harm during treatment. Further, when these rates are combined with no-change rates, only 40% or less of patients meaningfully recover. Importantly, treatment research has illuminated substantial variability in providers' outcomes. Simply put, the MHC provider impacts treatment outcomes, and stakeholders lack systematic access to valid and actionable information to optimize effective patient-provider matches. Without collecting and disseminating performance data, stakeholders lack vital information on which to base health care choices and personalize treatment. Conversely, there potentially is immense advantage to matching patients to providers based on scientific outcome data. Patients, stakeholders, researchers, and clinicians have all endorsed such applied knowledge transfer as a high priority. In response, the investigators have developed and piloted a technology to test this match concept and patient-centered health model.

Prominent health care agencies have placed outcome/performance measurement at the center of core initiatives. The Institute of Medicine specifically recommends integrating provider performance data in treatment decision-making. Despite this rhetoric, 2 Cochrane Reviews combined could only identify 4 studies that addressed this question with minimal methodology standards; the results were mixed. Importantly, none involved a targeted dissemination intervention, and none involved MHC. Previous research, including our own, has empirically demonstrated substantial differences in projected treatment effect sizes depending on to which therapist a patient is referred. The key evidence gap is the need for a rigorous test of the effectiveness of a targeted MHC provider-performance dissemination intervention compared to standard/pragmatic referral and case assignment. Relatedly, the Patient-Centered Outcomes Research Institute (PCORI) has called for increased "precision" or "personalized" treatment, with a focus on tailoring. The match algorithm responds directly to this high priority call to customize care in a personal and evidence-based way.

Specific Aims:

The aim of this comparative effectiveness research (CER) is to test an innovative, scientifically informed patient-therapist referral match algorithm based on MHC provider outcome data. The investigators will employ a randomized controlled trial (RCT) to compare the match algorithm with the commonplace pragmatic referral matching (based on provider availability, convenience, or self-reported specialty). Psychosocial treatment itself will remain naturalistically administered by varied providers (e.g., psychologists, social workers) to patients with complex mental health concerns within a partner clinic network, Psychological and Behavioral Consultants (PsychBC). The investigators hypothesize that the scientific match group will outperform the pragmatic match group in decreasing patient symptoms and treatment dropout, and in promoting patient functional outcomes, outcome expectations, and care satisfaction, as well as patient-therapist alliance quality. Doing so will establish the match algorithm as a mechanism of effective patient-centered MHC.

Methods:

The investigators will compare the effectiveness of naturalistic MHC either with or without the scientific matching aid with a double blind, individual level RCT. The investigators will first conduct a baseline assessment of PsychBC therapists' (target enrollment N=44) performance (across at least 15 cases) to determine their strengths in treating 12 behavioral health domains measured by the primary outcome tool on which our match algorithm is based -- the Treatment Outcome Package (TOP). The TOP is already administered routinely in our partner network. Based on years of predictive analytic research, this tool classifies therapists as "effective," "neutral," or "ineffective/harmful" for each TOP domain. The blinded therapists will be crossed over conditions.

Next, for the trial, new adult outpatients (target enrollment N=281) will be randomly assigned to the Match condition or case assignment as usual (typically based on pragmatic considerations, such as provider availability, convenience, or self-reported specialty). The only patient exclusion criterion will be people who are not the primary decision-maker for their care. Thus, patients will present with a multitude of problems across a spectrum of diagnoses. With therapist assignment as the only manipulation, participating therapists will treat patients fully naturalistically. Treatment outcomes will be assessed regularly through mutual termination or up to 16 weeks. Primary analyses will involve hierarchical linear modeling to examine comparative rates and patterns of change on the outcomes.

ELIGIBILITY:
Inclusion:

* Being 18-70 years of age
* Being the primary, informed decision-maker for one's care
* Willingness to be randomized to condition and to complete a few study-specific measures

Exclusion:

* Being under 18 or over 70 years of age
* Not being responsible for one's own treatment decisions
* Unwillingness to be randomized to condition and/or to complete a few study-specific measures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Constantino, PhD, Principal Investigator — University of Massachusetts, Amherst; James F Boswell, PhD, Principal Investigator — University at Albany, SUNY; David R Kraus, PhD, Principal Investigator — Outcome Referrals, Inc.; Thomas P Swales, PhD, Principal Investigator — Psychological and Behavioral Consultants
Locations (1):
- University of Massachusetts Amherst, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request on a case-by-case basis, we will share all IPD that underlie results in a publication (e.g., data extraction for meta-analyses). As appropriate, based on specific scientific journals' standards, we will provide analytic code used to generate published results.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We will begin sharing IPD upon request 6 months following the publication of our peer-reviewed final research report for PCORI, and we will maintain our de-identified data set indefinitely given possible future requests (e.g., to extract data for meta-analyses).
Access Criteria: We will share fully de-identified IPD, a corresponding data dictionary, and the above supporting information to professional scientific colleagues (with established reputations for publishing original psychotherapy research in accordance with ethical guidelines) for the purposes of replication efforts or meta-analyses. For other usages, such as requests to conduct novel secondary analyses, we will consider such collaborations on a case-by-case basis and clearly determine authorship arrangements in writing.
  Review requests, including a detailed plan for how the data will be used, should be directed via email to the PI, Dr. Michael Constantino (mconstantino@psych.umass.edu). Dr. Constantino reserves the right to deny individual share requests if the usage details are questionable or unclear.

REFERENCES:
- [Derived] Coyne AE, Gaines AN, DeFontes CG, Constantino MJ, Barcala-Delgado DI, Boswell JF, Kraus DR. Parsing the existential isolation-outcome association into its within- and between-patient components in naturalistic psychotherapy. Psychotherapy (Chic). 2025 Jun;62(2):235-242. doi: 10.1037/pst0000564. Epub 2025 Jan 20. PMID 39836135
- [Derived] Boswell JF, Constantino MJ, Coyne AE, Kraus DR. For whom does a match matter most? Patient-level moderators of evidence-based patient-therapist matching. J Consult Clin Psychol. 2022 Jan;90(1):61-74. doi: 10.1037/ccp0000644. Epub 2021 Jun 10. PMID 34110861
- [Derived] Constantino MJ, Boswell JF, Coyne AE, Swales TP, Kraus DR. Effect of Matching Therapists to Patients vs Assignment as Usual on Adult Psychotherapy Outcomes: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Sep 1;78(9):960-969. doi: 10.1001/jamapsychiatry.2021.1221. PMID 34106240
- See also: Study-specific website — http://improvementalhealthcare.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pragmatic Match | Scientific Match
Started | 155 (155 patients were randomly assigned to the Pragmatic Match condition) | 133 (133 patients were randomly assigned to the Scientific Match condition)
Begin Treatment | 119 (119 Pragmatic Match patients actually began treatment (attended at least 1 session)) | 99 (99 Scientifically Matched patients actually began treatment (attended at least one session))
Completed | 119 (119 patients provided naturalistic treatment data and were included in analyses) | 99 (99 patients provided naturalistic treatment data and were included in analyses)
Not Completed | 36 | 34
Not completed — Failed to provide data beyond baseline | 36 | 34

BASELINE CHARACTERISTICS:
Population: Baseline analysis population N = 218, or the final analysis sample of patients who attended at least one treatment session
Groups:
- Total: Total of all reporting groups
Arm/Group | Pragmatic Match | Scientific Match | Total
Number analyzed (Participants) | 119 | 99 | 218
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 119 | 99 | 218
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.42 (11.55) | 33.33 (10.72) | 33.93 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 66 | 147
  Male | 38 | 33 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 116 | 96 | 212
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 106 | 87 | 193
  Hispanic or Latino | 3 | 3 | 6
  African American/Black | 6 | 7 | 13
  American Indian or Alaska Native | 0 | 0 | 0
  East Indian | 0 | 1 | 1
  Other | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 119 | 99 | 218
Treatment Outcome Package-Clinical Scales (TOP-CS): General Impairment [Mean (Standard Deviation); unit: units on a scale] — The TOP-CS consists of 58 items assessing 12 symptom/functional domains: depression, quality of life, mania, panic, psychosis, substance abuse, social conflict, sexual functioning, sleep, suicidality, violence, and work functioning. The items are used to create domain-specific z-scores that reflect SDs relative to the general population mean. To create an index of global impairment, the 12 domain-specific z-scores are averaged. Higher scores represent greater impairment (e.g., 0 represents the general population mean, +2 represents impairment that is 2 SDs above the population mean).
  units on a scale | 0.86 (0.78) | 1.04 (.96) | 0.94 (0.87)
Symptom Checklist-10 (SCL-10): Global Psychological Distress [Mean (Standard Deviation); unit: units on a scale] — The Symptom Checklist-10 (SCL-10) was used to assess global psychological distress. The 10 items are rated from 0-4 and summed to create a total score (theoretical range = 0-40), with higher scores indicating greater distress.
  units on a scale | 15.48 (7.93) | 16.08 (7.74) | 15.75 (7.83)

OUTCOME MEASURES:

1. Primary Outcome: Average Z-Scores for the Treatment Outcome Package-Clinical Scales (TOP-CS; Kraus, Seligman, & Jordan, 2005)
Description: The TOP-Clinical Scales consist of 58 items assessing 12 symptom and functional domains (risk-adjusted for case mix variables assessed via 37 items on the companion TOP-Case Mix form, such as divorce, job loss, comorbidity): work functioning, sexual functioning, social conflict, depression, panic/somatic anxiety, psychosis, suicidal ideation, violence, mania, sleep, substance abuse, and quality of life. Global symptom severity was assessed by averaging the z-scores (i.e., standard deviation units relative to the general population mean) across the 12 clinical scales. Higher scores indicate greater impairment. Given that we examined change over the entire treatment period for this outcome (in a longitudinal hierarchical linear model), we provide the average mean and standard deviation for the TOP-CS z-scores across all measurement occasions.
Time Frame: Baseline and biweekly across 16 weeks
Population: All participants who were randomized to condition and completed at least one assessment after baseline (N = 218)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pragmatic Match | Scientific Match
Number analyzed (Participants) | 119 | 99
units on a scale | 0.57 (0.80) | 0.56 (0.82)
Statistical Analysis 1: Comparison: Pragmatic Match vs Scientific Match; To account for the nested nature of the data (time points nested within patients nested within therapists), a 3-level hierarchical linear model was used to test the effect of condition (Scientific Match = 1; Pragmatic Match = 0) on weekly during-treatment change on the TOP-CS average z-scores. Given that higher TOP-CS z-scores indicate greater impairment, negative slopes indicate a weekly decrease in impairment during treatment (i.e., a better outcome or more improvement); Test type: Superiority — We used the Optimal Design program to determine the minimum numbers of therapists and patients needed to detect a moderate effect of condition (standardized difference between change rates = .50). Based on this a priori power analysis, we will need a total of 44 therapists and 211 patients to achieve a power of .80 to detect moderate condition effects. Factoring in a 25% dropout rate, enrolling 281 patients should provide sufficient statistical power; p = .02, 3-level hierarchical linear model; condition effect on weekly change rate = -0.04, 95% CI 2-sided [-0.05 to -0.03], Standard Error of Mean 0.01

2. Secondary Outcome: Symptom Checklist-10 (SCL-10; Rosen, Drescher, Moos, & Gusman, 1999) Total Score
Description: Global psychological distress was assessed with the Symptom Checklist-10 (SCL-10; Rosen, Drescher, Moos, & Gusman, 1999), a 10-item, well validated and widely used self-report inventory that assesses psychological well-being. Total scores can range from 0 to 40, with higher scores indicating greater distress. Given that we examined change over the entire treatment period for this outcome (in a longitudinal hierarchical linear model), we provide the average mean and standard deviation for the SCL-10 total score across all measurement occasions.
Time Frame: Baseline and biweekly across 16 weeks
Population: All participants who were randomized to condition and completed at least one assessment after baseline (N = 218)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pragmatic Match | Scientific Match
Number analyzed (Participants) | 119 | 99
units on a scale | 12.52 (8.01) | 12.06 (7.70)
Statistical Analysis 1: Comparison: Pragmatic Match vs Scientific Match; To account for the nested nature of the data (time points nested within patients nested within therapists), a 3-level hierarchical linear model was used to test the effect of condition (Scientific Match = 1; Pragmatic Match = 0) on weekly during-treatment change on the SCL-10 total score. Given that higher SCL-10 scores indicate greater psychological distress, negative slopes indicate a weekly decrease in impairment during treatment (i.e., a better outcome or more improvement); Test type: Superiority; p = .03, 3-level hierarchical linear model; condition effect on weekly change rate = -0.16, 95% CI 2-sided [-0.30 to -0.02], Standard Error of Mean 0.07

3. Secondary Outcome: Working Alliance Inventory-Short Form, Patient Version (WAI-SF-P; Tracey, & Kokotovic, 1989) Total Score
Description: The WAI is the most widely used alliance measure, assessing patient-therapist agreement on the goals and tasks of treatment, and the quality of their relational bond. This 12-item short form assesses these dimensions from the patient's perspective, with higher scores indicating a more positive relationship (theoretical range = 12 to 84). Given that we examined change over the entire treatment period for this outcome (in a longitudinal hierarchical linear model), we provide the average mean and standard deviation for the WAI total score across all measurement occasions.
Time Frame: Biweekly across 16 weeks
Population: All participants who were randomized to condition and completed at least one assessment after baseline (N = 218)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pragmatic Match | Scientific Match
Number analyzed (Participants) | 119 | 99
units on a scale | 66.75 (13.35) | 68.44 (12.00)
Statistical Analysis 1: Comparison: Pragmatic Match vs Scientific Match; To account for the nested nature of the data (time points nested within patients nested within therapists), a 3-level hierarchical linear model was used to test the effect of condition (Scientific Match = 1; Pragmatic Match = 0) on weekly during-treatment change on the patient-rated WAI. Given that higher WAI scores indicate better quality therapeutic alliances, positive slopes indicate a weekly increase in alliance during treatment (i.e., a better outcome or more improvement); Test type: Superiority; p = .65, 3-level hierarchical linear model; condition effect on weekly change rate = -0.07, 95% CI 2-sided [-0.33 to 0.21], Standard Error of Mean 0.15

4. Secondary Outcome: Outcome Expectation (OE) Subscale of the Credibility/Expectancy Scale (CEQ; Devilly, & Borkovec, 2000)
Description: The OE subscale of the CEQ is the most widely used and psychometrically sound measure of patients' expectations for the personal efficacy of treatment. The three OE items range from 1-9 or 0-100% (in 10 percentage point increments), with higher ratings indicating greater expectation for improvement. Given that the OE CEQ items are assessed on different scales, we re-scaled the items to the same metric before creating a total score (theoretical range = 3 to 27). Given that we examined change over the entire treatment period for this outcome (in a longitudinal hierarchical linear model), we provide the average mean and standard deviation for the OE subscale across all measurement occasions.
Time Frame: Biweekly across 16 weeks
Population: All participants who were randomized to condition and completed at least one assessment after baseline (N = 218)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pragmatic Match | Scientific Match
Number analyzed (Participants) | 119 | 99
units on a scale | 18.12 (5.45) | 19.15 (5.30)
Statistical Analysis 1: Comparison: Pragmatic Match vs Scientific Match; To account for the nested nature of the data (time points nested within patients nested within therapists), a 3-level hierarchical linear model was used to test the effect of condition (Scientific Match = 1; Pragmatic Match = 0) on weekly during-treatment change on the OE subscale of the CEQ. Given that higher OE scores indicate more optimistic expectations, positive slopes indicate a weekly increase in OE during treatment (i.e., a better outcome or more improvement); Test type: Superiority; p = .41, 3-level hierarchical linear model; condition effect on weekly change rate = -0.06, 95% CI 2-sided [-0.17 to 0.07], Standard Error of Mean 0.07

5. Secondary Outcome: Domain-Specific Impairment on the Most Elevated Domain of the Treatment Outcome Package-Clinical Scales (TOP-CS)
Description: The TOP-CS consists of 58 items assessing 12 symptom and functional domains (risk-adjusted for case mix variables assessed via 37 items on the companion TOP-Case Mix form, such as divorce, job loss, comorbidity): work functioning, sexual functioning, social conflict, depression, panic/somatic anxiety, psychosis, suicidal ideation, violence, mania, sleep, substance abuse, and quality of life. Domain-specific impairment reflects each patient's scores on their most elevated problem domain (i.e., the domain most elevated at baseline). These scores were standardized z-scores (i.e., standard deviation units relative to the general population mean), with higher scores indicating greater impairment. Given that we examined change over the treatment period for this outcome (hierarchical linear model), we provide the average mean and standard deviation for the most elevated TOP domain across all measurement occasions. Note that this measure was positively skewed so we log-transformed it.
Time Frame: Baseline and biweekly across 16 weeks
Population: All participants who were randomized to condition and completed at least one assessment after baseline (N = 218)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pragmatic Match | Scientific Match
Number analyzed (Participants) | 119 | 99
units on a scale | 0.27 (.24) | 0.28 (0.23)
Statistical Analysis 1: Comparison: Pragmatic Match vs Scientific Match; To account for the nested nature of the data (time points nested within patients nested within therapists), a 3-level hierarchical linear model was used to test the effect of condition (Scientific Match = 1; Pragmatic Match = 0) on weekly during-treatment change on the log-transformed TOP-CS domain-specific z-scores. Given that higher z-scores indicate greater impairment, negative slopes indicate a weekly decrease in impairment during treatment (i.e., a better outcome or more improvement); Test type: Superiority; p = .01, 3-level hierarchical linear model; condition effect on weekly change rate = -0.01, 95% CI 2-sided [-0.01 to -0.006], Standard Error of Mean 0.002

6. Secondary Outcome: Early Treatment Discontinuation (i.e., Attending 2 or Fewer Treatment Sessions)
Description: Early treatment discontinuation was operationalized as a patient discontinuing treatment after 2 or fewer sessions, whereas early continuation was operationalized as attending 3 or more treatment sessions. For analyses, early treatment discontinuation was coded 1 and early continuation was coded 0.
Time Frame: Early treatment discontinuation/continuation at session 2
Population: All participants who were randomized to condition and completed at least one assessment after baseline (N = 218)
Measure: Count of Participants; unit: Participants
Arm/Group | Pragmatic Match | Scientific Match
Number analyzed (Participants) | 119 | 99
Participants | 22 | 22
Statistical Analysis 1: Comparison: Pragmatic Match vs Scientific Match; Multilevel logistic regression analysis with patients nested within therapists (Scientific Match = 1; Pragmatic Match = 0). Statistically significant odds ratios that are greater than 1 would indicate that patients in the Scientific Match Condition were more likely to discontinue treatment early, whereas odds ratios that are less than 1 would indicate the opposite; Test type: Superiority; p = .48, Multilevel logistic regression; Odds Ratio (OR) = 1.30, Standard Error of Mean 0.48

7. Secondary Outcome: Overall Provider Quality Subscale of the Treatment Outcome Package (TOP) Satisfaction Scale
Description: The Overall Provider Quality subscale of the TOP Satisfaction Scale assesses the extent to which patients are satisfied with their mental health care provider. This subscale reflects the average of 4 items, with higher scores indicating greater satisfaction (theoretical range = 1 to 6).
Time Frame: Assessed after 16 weeks of treatment or at the point of naturalistic treatment termination, whichever comes sooner
Population: Due to a relatively large amount of missing data for this measure (compared to other study measures), this was considered a completer analysis that involved only the patients who completed this posttreatment measure (N = 97).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pragmatic Match | Scientific Match
Number analyzed (Participants) | 54 | 43
units on a scale | 5.01 (1.35) | 5.17 (1.11)
Statistical Analysis 1: Comparison: Pragmatic Match vs Scientific Match; Due to the nested nature of the data (patients nested within therapists), we used a two-level hierarchical linear model to test the effect of condition on provider satisfaction at posttreatment. Because higher values indicate more satisfaction, a positive condition effect would indicate that Scientific Match patients were more satisfied than Pragmatic Match patients, whereas a negative condition effect would indicate the opposite; Test type: Superiority; p = .44, 2-level hierarchical linear model; condition effect on satisfaction = 0.37, 95% CI 2-sided [-0.57 to 1.31], Standard Error of Mean 0.48

ADVERSE EVENTS:
Time Frame: Psychotherapy was delivered naturalistically. Therefore, treatment lengths varied. Patients completed study measures through the point of actual treatment termination or through 16 weeks of treatment (whichever came sooner).
Arm/Group | Pragmatic Match | Scientific Match
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/99
Other Adverse Events (participants affected / at risk) | 0/119 | 0/99

LIMITATIONS AND CAVEATS:
The naturalistic design resulted in limited information on the treatments themselves, differing treatment lengths, and some missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/00/NCT02990000/Prot_SAP_ICF_000.pdf